CLINICAL TRIAL: NCT04124900
Title: Measurement of Telomere Associated Variables (TAVs) for Diagnostic Purposes in Prostate Cancer
Brief Title: Telomere Associated Variables (TAVs) in Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Life Length SL (Industry)
Responsible Party: Sponsor
Other Study IDs: PROSTAV001
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostate biopsy; telomere; biomarker; screening; prostate; cancer; biopsy
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMCs isolated from fresh blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients at prostate cancer risk diagnosed: The study is composed of one single subject cohort. After risk evaluation, prostate biopsies will be performed for diagnostic purposes on all recruited patients. The cases are sorted into two groups after diagnosis:
  * Group 1: patients at prostate cancer risk diagnosed with significant prostate cancer after prostatic biopsy (Gleason >6).
  * Group 2: patients at prostate cancer risk diagnosed free of cancer after prostate biopsy. There will be a subdivision within this group in patients without significant prostate cancer ( No cancer o Non-significant prostate cancer (Gleason ≤6)).

SUMMARY:
This research project results from the interest in continuing the collaboration with the previous LL-HURS-ONC001 clinical validation study, which gives cause to the present study. LL-HURS-ONC001 was carried out with the participation of HURS' Principal Investigator and the team of experts in prostate cancer, as well as with the participation of the Sponsor's scientific and development team, Life Length SL, led by Dr. Najarro.

The main objective of this study is to demonstrate the efficacy of the PROSTAV test in cutting down on unnecessary biopsies in prostate cancer screening/early diagnosis. PROSTAV is a minimally invasive test, easy to implement as biomarker for prostate cancer diagnosis. The efficacy of the PROSTAV test is clinically validated by the results obtained in a previous study, LL-HURS-ONC001.

The purpose of this study is to advance in the development of new biomarkers in areas where there is a clinical need and where the telomeric profile influences medical decisions within the patient's clinical context. The association level between each individual's telomere biology and the results of the prostate biopsy will be confirmed. Data will be collected to subsequently delve deeper into and accurately establish the effect of this measure in prostate cancer patient management to substantiate its implementation in standard care.

DETAILED DESCRIPTION:
In this study, patient inclusion and sample collection are multicentric. Sample analysis will be carried out at Life Length's laboratories at the Madrid Science Park in Canto Blanco university campus.

The study will be initiated immediately after approval by the IRB and has an overall length of 12 months (recruiting time).

The main purpose of the present study is to determine the efficacy of the PROSTAV test as a prostate cancer biomarker developed by Life Length and which has been subject to internal validation in a previous study (LL-HURS-ONC001). For this purpose, the risk-prediction algorithm based on telomere and clinical variables will be used. This allows to back medical decisions in patients with uncertain PC diagnosis based on their PSA levels and the need to perform a prostate biopsy. The standard of care of the participating hospitals and following the European Urology Association recommendations, patients with PSA >3 (prostate-specific antigen) and/or positive digital rectal examination (DRE) are considered at risk for developing PC. However, some medical advisors of the sponsor stated that sometimes patients with PSA levels<3 are also diagnosed with prostate cancer. For this reason, it has been decided to remove the lower limit of PSA as inclusion criteria.

This study includes only one group of patients defined by inclusion criteria and who will be classified in different groups after a biopsy is performed: 1) patients with a positive biopsy result (diagnosed with significant prostate cancer) (Gleason score >6), and without significant prostate cancer (Gleason score ≤6) or no cancer. Before knowing the histopathological results of the biopsy, the PROSTAV test will be performed. Depending on the results of the PROSTAV test, the physician will write down which decision he or she would have made as to performing or not a biopsy: zero (0) for a low-risk result in the PROSTAV test, in which case no biopsy would have been performed; and one (1) for a PC risk result in the PROSTAV test, in which case a biopsy would have been performed. Regardless of what the result of the PROSTAV test is, all patients will undergo a biopsy since the result in PROSTAV test will not influence the standard of care in this study.

A 10 ml. sample is required from all subjects included in the study for telomere analysis. This sample is obtained from blood drawn before performing the diagnostic prostate biopsy. The sample must be drawn within a 90-day period prior to biopsy.

The design of the present project allows for one single study phase. This study is a clinical efficacy validation study in patients in whom the results of potential biopsy sparing are compared after evaluating medical decisions based on the use of the PROSTAV test.

The point of origin of the samples are the different participating centers that will use the samples for application of the telomere biology evaluation techniques.

Mononuclear cells in peripheral blood from all samples will be isolated and analyzed to determine values of Telomere Associated Variables (TAVs).

For the calculation of the telomere variables, the Sponsor will use the High-Throughput Quantitative Fluorescent in Situ Hybridization technique (HT-Q-FISH).

Data resulting from each biological sample will be analyzed to obtain a defined risk assessment based on the algorithm of the PROSTAV test. The purpose of the analysis is the integration of the data resulting from telomere measurements (average, median, percentage of short telomeres, ratio of short and long telomeres, etc.) and PSA and free PSA levels, age and the DRE results of the patient's medical record to determine whether they are low-risk patients, in which a biopsy would not be necessary to confirm presence of prostate cancer. By doing this, it is intending to demonstrate the efficacy of the PROSTAV test, since biopsies would be performed in any case and also show the test's sensitivity and specificity values in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* To be over 18 years of age.
* To have given written consent to participate in the study.
* To be classified as a patient at prostate cancer risk according to criteria of high PSA levels (<10 ng/ml) and the urologist's decision to perform a prostate biopsy in standard of care.
* To be diagnosed by a prostate biopsy with or without concomitant MRI.
* Caucasic race

Exclusion Criteria:

* Patients that have received Alpha-5 reductase therapy.
* Existing serious active liver, lung or kidney disease, as well as severe active infections.
* Existing serious disease or psychiatric disorder that prevents them from expressing informed consent and/or if patients are not able to follow protocol procedures and give their informed consent.
* Patients at risk resulting from conventional blood extraction.
* Subjects with active neoplasm diagnosed during the past five years.

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: The study population will include cases with high PSA levels (PSA<10 ng/ml) and with indication criterion for prostate cancer biopsy based on prostate cancer risk-related endpoints.
  The study is composed of one single subject cohort. After risk evaluation, prostate biopsies will be performed for diagnostic purposes on all recruited patients. The cases are sorted into two groups after diagnosis:
  * Group 1: patients at prostate cancer risk diagnosed with significant prostate cancer after prostatic biopsy (Gleason >6).
  * Group 2: patients at prostate cancer risk diagnosed free of cancer after prostate biopsy. There will be a subdivision within this group in patients without significant prostate cancer:
    * No cancer
    * Non-significant prostate cancer (Gleason ≤6).
Sampling Method: Non-Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Telomere Associated Variables | One day single measurement
  This is a clinical multicenter study focused on evaluating the efficacy of the PROSTAV test in patients at risk of prostate cancer based on data of telomere associated variables (TAV) as risk-score. The study comprises one single prospective observational phase.

CONTACTS AND LOCATIONS:
Overall Officials: Maria José Requena, Principal Investigator — University Hospital Reina Sofía; Enrique Gómez, MD, Principal Investigator — University Hospital Reina Sofía
Locations (10):
- United States (2):
  - Urological Research Network, Corp., Hialeah, Florida
  - Houston Methodist Research Institute, Houston, Texas
- Spain (8):
  - Hospital Infanta Margarita, Cabra, Córdoba
  - Instituto Médico Tecnológico, Barcelona
  - University Hospital Reina Sofía, Córdoba
  - ROC Clinic, Madrid
  - Instituto de Urología LYX, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Doce de Octubre, Madrid
  - Instituto Valenciano de Oncología, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanahan D, Weinberg RA. The hallmarks of cancer. Cell. 2000 Jan 7;100(1):57-70. doi: 10.1016/s0092-8674(00)81683-9. No abstract available. PMID 10647931
- [Background] Shay JW, Wright WE, Werbin H. Defining the molecular mechanisms of human cell immortalization. Biochim Biophys Acta. 1991 Apr 16;1072(1):1-7. doi: 10.1016/0304-419x(91)90003-4. PMID 1850299
- [Background] Hahn WC, Counter CM, Lundberg AS, Beijersbergen RL, Brooks MW, Weinberg RA. Creation of human tumour cells with defined genetic elements. Nature. 1999 Jul 29;400(6743):464-8. doi: 10.1038/22780. PMID 10440377
- [Background] Wright WE, Shay JW. Telomere dynamics in cancer progression and prevention: fundamental differences in human and mouse telomere biology. Nat Med. 2000 Aug;6(8):849-51. doi: 10.1038/78592. PMID 10932210
- [Background] Shay JW, Zou Y, Hiyama E, Wright WE. Telomerase and cancer. Hum Mol Genet. 2001 Apr;10(7):677-85. doi: 10.1093/hmg/10.7.677. PMID 11257099
- [Background] Kim NW, Piatyszek MA, Prowse KR, Harley CB, West MD, Ho PL, Coviello GM, Wright WE, Weinrich SL, Shay JW. Specific association of human telomerase activity with immortal cells and cancer. Science. 1994 Dec 23;266(5193):2011-5. doi: 10.1126/science.7605428.
- [Background] Shay JW, Bacchetti S. A survey of telomerase activity in human cancer. Eur J Cancer. 1997 Apr;33(5):787-91. doi: 10.1016/S0959-8049(97)00062-2. PMID 9282118
- [Background] Breslow RA, Shay JW, Gazdar AF, Srivastava S. Telomerase and early detection of cancer: a National Cancer Institute workshop. J Natl Cancer Inst. 1997 May 7;89(9):618-23. doi: 10.1093/jnci/89.9.618. No abstract available. PMID 9150185
- [Background] Shay JW. Telomerase in cancer: diagnostic, prognostic, and therapeutic implications. Cancer J Sci Am. 1998 May;4 Suppl 1:S26-34. No abstract available. PMID 9619268
- [Background] Norton JC, Holt SE, Wright WE, Shay JW. Enhanced detection of human telomerase activity. DNA Cell Biol. 1998 Mar;17(3):217-9. doi: 10.1089/dna.1998.17.217. PMID 9539101
- [Background] Hiyama E, Hiyama K, Yokoyama T, Matsuura Y, Piatyszek MA, Shay JW. Correlating telomerase activity levels with human neuroblastoma outcomes. Nat Med. 1995 Mar;1(3):249-55. doi: 10.1038/nm0395-249. PMID 7585042
- [Background] Sommerfeld HJ, Meeker AK, Piatyszek MA, Bova GS, Shay JW, Coffey DS. Telomerase activity: a prevalent marker of malignant human prostate tissue. Cancer Res. 1996 Jan 1;56(1):218-22. PMID 8548767
- [Background] Mehle C, Piatyszek MA, Ljungberg B, Shay JW, Roos G. Telomerase activity in human renal cell carcinoma. Oncogene. 1996 Jul 4;13(1):161-6. PMID 8700542
- [Background] Tatsumoto N, Hiyama E, Murakami Y, Imamura Y, Shay JW, Matsuura Y, Yokoyama T. High telomerase activity is an independent prognostic indicator of poor outcome in colorectal cancer. Clin Cancer Res. 2000 Jul;6(7):2696-701. PMID 10914712
- [Background] Shay JW, Gazdar AF. Telomerase in the early detection of cancer. J Clin Pathol. 1997 Feb;50(2):106-9. doi: 10.1136/jcp.50.2.106. PMID 9155689
- [Background] Gurel B, Iwata T, Koh CM, Yegnasubramanian S, Nelson WG, De Marzo AM. Molecular alterations in prostate cancer as diagnostic, prognostic, and therapeutic targets. Adv Anat Pathol. 2008 Nov;15(6):319-31. doi: 10.1097/PAP.0b013e31818a5c19. PMID 18948763
- [Background] Heaphy CM, Meeker AK. The potential utility of telomere-related markers for cancer diagnosis. J Cell Mol Med. 2011 Jun;15(6):1227-38. doi: 10.1111/j.1582-4934.2011.01284.x. PMID 21352473
- [Background] Hou L, Joyce BT, Gao T, Liu L, Zheng Y, Penedo FJ, Liu S, Zhang W, Bergan R, Dai Q, Vokonas P, Hoxha M, Schwartz J, Baccarelli A. Blood Telomere Length Attrition and Cancer Development in the Normative Aging Study Cohort. EBioMedicine. 2015 Apr 13;2(6):591-6. doi: 10.1016/j.ebiom.2015.04.008. eCollection 2015 Jun. PMID 26288820
- [Background] Mottet N, Bellmunt J, Bolla M, Briers E, Cumberbatch MG, De Santis M, Fossati N, Gross T, Henry AM, Joniau S, Lam TB, Mason MD, Matveev VB, Moldovan PC, van den Bergh RCN, Van den Broeck T, van der Poel HG, van der Kwast TH, Rouviere O, Schoots IG, Wiegel T, Cornford P. EAU-ESTRO-SIOG Guidelines on Prostate Cancer. Part 1: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2017 Apr;71(4):618-629. doi: 10.1016/j.eururo.2016.08.003. Epub 2016 Aug 25. PMID 27568654
- [Background] Humphrey PA, Moch H, Cubilla AL, Ulbright TM, Reuter VE. The 2016 WHO Classification of Tumours of the Urinary System and Male Genital Organs-Part B: Prostate and Bladder Tumours. Eur Urol. 2016 Jul;70(1):106-119. doi: 10.1016/j.eururo.2016.02.028. Epub 2016 Mar 17. PMID 26996659
- See also: Requirements for Minimum Sample Size for Sensitivity and Specificity Analysis — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5121784/pdf/jcdr-10-YE01.pdf